CLINICAL TRIAL: NCT05806567
Title: A Three-part, Sequential, Non-randomized, Open-label Study Designed to Evaluate the Effect of Oral Belumosudil on UGT1A1, P-gp, BCRP and OATP1B1 Inhibition in the Fed State in Healthy Male Subjects
Brief Title: A Study to Assess the Effect of Oral Belumosudil on Inhibition of Various Proteins in the Fed State in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kadmon, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: INT17676; U1111-1277-6732 (Registry Identifier: ICTRP)
Record Dates: First submitted 2023-03-28; First posted 2023-04-10 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Immune System Disorder; Healthy Volunteers
MeSH Terms: conditions — Immune System Diseases | interventions — belumosudil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1 (Experimental): Belumosudil + UGT1A1 victim drug administered in the fed state
  Interventions: Drug: Belumosudil; Drug: UGT1A1 victim drug
- Part 2 (Experimental): Belumosudil + P-gp victim drug administered in the fed state
  Interventions: Drug: Belumosudil; Drug: P-gp victim drug
- Part 3 (Experimental): Belumosudil + OATP1B1/BCRP victim drug administered in the fed state
  Interventions: Drug: Belumosudil; Drug: OATP1B1/BCRP victim drug

INTERVENTIONS:
Drug: Belumosudil — Pharmaceutical form: Tablet; Route of administration: Oral
  Other Names: REZUROCK/KD025/SAR445761
Drug: UGT1A1 victim drug — Pharmaceutical form: Tablet; Route of administration: Oral
  Arms: Part 1
Drug: P-gp victim drug — Pharmaceutical form: Capsule; Route of administration: Oral
  Arms: Part 2
Drug: OATP1B1/BCRP victim drug — Pharmaceutical form: Tablet; Route of administration: Oral
  Arms: Part 3

SUMMARY:
The purpose of this study is to evaluate safety and pharmacokinetics (PK) effect of belumosudil on the uridine diphosphate glucuronosyltransferase (UGT)1A1 (Part 1), P glycoprotein (P-gp) (Part 2) and breast cancer resistance protein (BCRP)/organic anion transporting polypeptide (OATP)1B1 (Part 3) inhibition in the fed state in healthy male subjects.

DETAILED DESCRIPTION:
Part 1: The estimated time from screening until the follow-up phone call is approximately 6 weeks per subject.

Part 2: The estimated time from screening until the follow-up phone call is approximately 7 weeks per subject.

Part 3: The estimated time from screening until the follow-up phone call is approximately 7 weeks per subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male participants aged 18 to 55 years old
* Must agree to use an adequate method of contraception
* Must be able to understand and provide a written informed consent

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients.
* Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hay fever is allowed unless it is active.
* Significant serious skin disease, including rash, food allergy, eczema, psoriasis, or urticaria.
* Failure to satisfy the investigator of fitness to participate for any other reason.

The above information is not intended to contain all considerations relevant to the potential participation in a clinical trial.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2022-07-27 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2022-10-28 (Actual)

PRIMARY OUTCOMES:
AUC(0-last)- Parts 1,2, and 3 (victim drugs) | Multiple timepoints up to approximately 15 days
  Area under the curve from time 0 to the time of last measurable concentration
AUC(0-inf)- Parts 1,2, and 3 (victim drugs | Multiple timepoints up to approximately 15 days
  Area under the curve from time 0 extrapolated to infinity

SECONDARY OUTCOMES:
Tmax- Parts 1, 2, and 3 (victim drugs, belumosudil and belumosudil metabolites) | Multiple timepoints up to approximately 15 days
  Time of maximum observed concentration.
Cmax -Parts 1, 2, and 3 (victim drugs, belumosudil and belumosudil metabolites) | Multiple timepoints up to approximately 15 days
  Maximum observed concentration
T1/2 -Parts 1, 2, and 3 (victim drugs, belumosudil and belumosudil metabolites) | Multiple timepoints up to approximately 15 days
  Terminal elimination half-life
AUC(0-last)-Part 1 (victim metabolite) | Multiple timepoints up to approximately 10 days
AUC(0-inf)- Part 1 (metabolite of victim drug) | Multiple timepoints up to approximately 10 days
Tmax- Part 1(metabolite of victim drug) | Multiple timepoints up to approximately 10 days
Cmax- Part 1 (metabolite of victim drug) | Multiple timepoints up to approximately 10 days
T1/2- Part 1 (metabolite of victim drug) | Multiple timepoints up to approximately 10 days
AUC(0-last) - Parts 1, 2, and 3 (Belumosudil and metabolites) | Multiple timepoints up to approximately 15 days
Area under the curve for the defined interval between doses (tau) [AUC(0 tau)] - Parts 1, 2, and 3 | Multiple timepoints up to approximately 15 days
  Area under the curve for the defined interval between doses (tau)
Number of participants with adverse events (AEs) and serious adverse events (SAEs) | Up to 30 days after the administration of last dose of study drug i.e., up to approximately 43 days
  To provide additional safety and tolerability information for belumosudil by assessing: AEs, vital signs, ECGs, physical examinations and laboratory safety tests following administration of the three victim drugs alone and in combination with belumosudil.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number: 8400001, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: INT17676 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25274&tenant=MT_SNY_9011